CLINICAL TRIAL: NCT06824987
Title: Phase 2b Multicentre, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Dose-Ranging Study to Assess the Efficacy, Safety, and Tolerability of AZD2373 in Participants With APOL1-Mediated Kidney Disease (APPRECIATE)
Brief Title: Dose-Ranging Safety, Tolerability, and Efficacy Study of AZD2373 in Participants With APOL1-Mediated Kidney Disease
Acronym: APPRECIATE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6800C00005
Record Dates: First submitted 2025-01-24; First posted 2025-02-13 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: APOL1-Mediated Kidney Disease
Keywords: APOL1-Mediated Kidney Disease; AZD2373

STUDY DESIGN:
Intervention Model Description: Participants will be randomized at a 1:1:1 ratio to 3 study treatment arms:
  * Placebo group
  * AZD2373 - Arm 1
  * AZD2373 - Arm 2
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: AZD2373 (study drug) and placebo will be provided in identical Accessorized pre-filled glass syringes.
  The Interactive Response technology / Randomisation and Trial Supply Management (IRT/RTSM) will provide to the investigator(s) or pharmacists the kit identification number to be allocated to the participant at the dispensing visit.
  Routines for this will be described in the IRT/RTSM user manual provided to each centre.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (3):
- Placebo group (Placebo Comparator): Participants will be randomized at a 1:1:1 ratio to 3 study treatment arms. Participants will receive SC injection of the assigned dose.
  Interventions: Combination Product: Placebo; Device: APOL1 Genotyping Clinical Trial Assay
- AZD2373 - Arm 1 (Experimental): Participants will be randomized at a 1:1:1 ratio to 3 study treatment arms. Participants will receive SC injection of the assigned dose.
  Interventions: Combination Product: AZD2373-Arm 1; Device: APOL1 Genotyping Clinical Trial Assay
- AZD2373 - Arm 2 (Experimental): Participants will be randomized at a 1:1:1 ratio to 3 study treatment arms. Participants will receive SC injection of the assigned dose.
  Interventions: Combination Product: AZD2373-Arm 2; Device: APOL1 Genotyping Clinical Trial Assay

INTERVENTIONS:
Combination Product: AZD2373-Arm 1 — Accessorized Pre-Filled Syringe (Solution for injection)
  Arms: AZD2373 - Arm 1
Combination Product: AZD2373-Arm 2 — Accessorized Pre-Filled Syringe (Solution for injection)
  Arms: AZD2373 - Arm 2
Combination Product: Placebo — Accessorized Pre-Filled Syringe (Solution for injection).
  Arms: Placebo group
Device: APOL1 Genotyping Clinical Trial Assay — The APOL1 Genotyping Clinical Trial Assay, an investigational use only qualitative Polymerase Chain Reaction invitro diagnostic assay, discriminates between the rs73885319 G1(S342G) and rs71785313 G2 genotypes within the APOL1 gene from DNA extracted from whole blood.

SUMMARY:
The purpose of this study is to assess the efficacy and safety of AZD2373 in participants diagnosed with APOL1-Mediated Kidney Disease (AMKD) who are homozygotes or compound heterozygotes for APOL1 high-risk genotypes (G1 and G2). The primary hypothesis to be evaluated is that AZD2373, compared with placebo, will result in a greater reduction in UACR as assessed by the relative change from Baseline in UACR at Week 30.

DETAILED DESCRIPTION:
This is a Phase 2b study to assess efficacy and safety of AZD2373 involving 3 study treatment arms where participants and study personnel including study investigators are blinded to the assigned treatment.

Participants with 300 mg/g or greater UACR and eGFR ≥ 25mL/min/1.73m2 will be recruited into the study. Participants on kidney replacement therapy (dialysis or kidney transplant) or any other organ transplant will be excluded.

All participants will remain in the study on treatment until the last participant has completed 30 weeks of treatment. The treatment duration will be up to minimum of 30 weeks of study treatment.

Approximately 96 participants will be randomized to study intervention (approximately 32 participants in each treatment group).

ELIGIBILITY:
Inclusion Criteria:

* Age: Male and female participants aged 18 to 65 years, inclusive at the time of informed consent.
* Participants who have high-risk APOL1 genotype (G1/G1; G1/G2; G2/G2). The screening period can be extended if there are delays related to the shipment, handling, or processing of genotype results.
* A geometric mean UACR ≥ 300 mg/g calculated based on the mean of readings taken from 3 FMV urine samples collected on 3 consecutive days. Since the mean will be assessed for eligibility, any of the 3 readings may fall below 300 mg/g.
* eGFR ≥ 25 mL/min/1.73m2.
* Contraceptive use by males or females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

* Participants with diagnosis of Type 1 diabetes mellitus.
* Body Mass Index > 45 kg/m2.
* SBP > 180 mmHg/DBP > 110 mmHg (measured when the participant is considered to be at steady state, and preferably when they have taken their BP medications that same day).
* QTcF > 470 ms.
* Acute coronary syndrome/Acute myocardial infraction +/- coronary intervention with Percutaneous coronary intervention or Coronary artery bypass grafting within 6 months.
* Transient ischaemic attack/ stroke within 3 months.
* High second to third degree AV block or clinically significant sinus node dysfunction untreated with pacemaker.
* A history of ventricular arrhythmias requiring treatment.
* Participants with Type 2 diabetes mellitus must be excluded if ANY of the following conditions are present:

  1. Current or any past use of insulin
  2. Screening Haemoglobin A1c > 8.0%
  3. Receiving more than one oral anti-hyperglycaemic agent (excluding SGLT inhibitors which can be taken in addition to one other oral anti-hyperglycaemic agent).
* Participant on kidney replacement therapy (dialysis or kidney transplant) or any other organ transplant.
* History or serologic evidence of autoimmune-mediated glomerular disease including but not limited to: lupus nephritis (positive lupus serology), ANCA associated vasculitis (antineutrophil cytoplasmic antibody), membranous nephropathy (anti-phospholipase A2 receptor antibody or other autoantibody associated with membranous nephropathy), anti-GBM disease (anti-GBM antibody), or IgA nephropathy.
* Another underlying cause of kidney disease that is not associated with APOL1, including but not limited to polycystic kidney disease or, congenital anomalies of the kidney and urinary tract.
* History of a diagnosed coagulopathy, a major unexplained bleeding event, or other high-risk bleeding diathesis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Relative change in Urine Albumin-Creatinine Ratio (UACR) | From Baseline at Week 30
  To assess the effect of AZD2373 versus placebo in reducing albuminuria

SECONDARY OUTCOMES:
Relative change in Urine Albumin-Creatinine Ratio (UACR) | From Baseline at the End of Treatment (Until the last participant completes Week 30)
  To assess the effect of AZD2373 versus placebo in reducing albuminuria
Relative change in Urine Protein-Creatinine Ratio (UPCR) | From Baseline at Week 30
  To assess the effect of AZD2373 versus placebo in reducing proteinuria
Relative change in Urine Protein-Creatinine Ratio (UPCR) | From Baseline at the End of Treatment (Until the last participant completes Week 30)
  To assess the effect of AZD2373 versus placebo in reducing proteinuria
Proportion of participants achieving a 45% or greater reduction in Urine Albumin-Creatinine Ratio (UACR) | From Baseline at Week 30
  To assess the proportion of participants achieving a 45% or greater Urine Albumin-Creatinine Ratio (UACR) reduction by treatment
Proportion of participants achieving a 45% or greater reduction in Urine Albumin-Creatinine Ratio (UACR) | From Baseline at the End of Treatment (Until the last participant completes Week 30)
  To assess the proportion of participants achieving a 45% or greater Urine Albumin-Creatinine Ratio (UACR) reduction by treatment
Relative change in eGFR | From Baseline at the End of Treatment (Until the last participant completes Week 30)
  To assess pooled AZD2373 doses versus placebo on eGFR change
Incidence of development of ADA and ADA titer (if participants are ADA-positive) | During treatment (up to Week 30) and follow-up (up to 12 weeks)
  To evaluate the immunogenicity of AZD2373
Plasma concentration | From Baseline at the End of Treatment (Until the last participant completes Week 30)
  To evaluate the PK of AZD2373
Adverse Events (AEs), Serious Adverse Events (SAEs), and Drug Adverse Events (DAEs). | From baseline at the End of Treatment (Until the last participant completes Week 30)
  To assess the safety and tolerability of ranging doses of AZD2373. These events will be collected according to the timepoints specified in the schedule of assessments, starting from the time of signing the Informed Consent Form (ICF).

CONTACTS AND LOCATIONS:
Locations (65):
- United States (60):
  - Research Site, Alabaster, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Irondale, Alabama
  - Research Site, Beverly Hills, California
  - Research Site, Gardena, California
  - Research Site, Los Angeles, California
  - Research Site, Valencia, California
  - Research Site, Brandon, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Pompano Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, Duluth, Georgia
  - Research Site, Hinesville, Georgia
  - Research Site, Lawrenceville, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Stockbridge, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Hinsdale, Illinois
  - Research Site, Lafayette, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Bethesda, Maryland
  - Research Site, Potomac, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Roseville, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Tupelo, Mississippi
  - Research Site, Brooklyn, New York
  - Research Site, Laurelton, New York
  - Research Site, New York, New York
  - Research Site, Cary, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Fayetteville, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Jacksonville, North Carolina
  - Research Site, Kinston, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, Columbia, South Carolina
  - Research Site, Orangeburg, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Conroe, Texas
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Mesquite, Texas
  - Research Site, Pearland, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Alexandria, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia
- United Kingdom (5):
  - Research Site, Birmingham
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/